CLINICAL TRIAL: NCT04813510
Title: Effect of Electroacupuncture on SAP With MODS: a Prospective, Double-blind, Randomized Controlled Trial
Brief Title: Effect of Electroacupuncture on SAP With MODS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jianbo Yu (Other)
Responsible Party: Sponsor-Investigator, Jianbo Yu, Department of Anesthesiology, Director, Chief physician, Professor, Doctoral tutor, Tianjin Nankai Hospital
Organization: Tianjin Nankai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EA-SAP-202103
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Severe Acute Pancreatitis
Keywords: Severe Acute Pancreatitis; Multiple Organ Disfunction Syndrome
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electroacupuncture treatment (Experimental): Participants in the treatment group underwent 30 minutes acupuncture (0.30mm×70mm) at Zusanli(ST36), Xiajuxu(ST39), Hegu(LI4), Neiguan(PC6) once a day for seven days. After"Deqi",electroacupuncture stimulation apparatus (HANS G6805-2, Huayi Co, Shanghai, China) isconnected and maintained the end of treatment.
  Interventions: Device: electroacupuncture treatment
- sham electroacupuncture treatment (Sham Comparator): Participants in the control group received shallow needling (0.30mm×25mm) at nonacupoints (located 1 inch beside acupoints). Specifically, the depth of needle insertion into nonacupoints is 3-5mm and avoided manual stimulation and no "Deqi" without actual current output.
  Interventions: Device: sham electroacupuncture treatment

INTERVENTIONS:
Device: electroacupuncture treatment — Participants in the treatment group underwent 60 minutes acupuncture (0.30mm×70mm) at Zusanli(ST36), Xiajuxu(ST39), Hegu(LI4), Neiguan(PC6) once a day for seven days. After"Deqi", electroacupuncture stimulation apparatus(HANS G6805-2, Huayi Co, Shanghai, China) is connected with the density wave (2/100 Hz), width 0.25 ms, intensity of 1 ~ 30 mA (gradually increase to the patient's maximum tolerance) and maintained the end of treatment.
  Arms: electroacupuncture treatment
Device: sham electroacupuncture treatment — Participants in the sham electroacupuncture group received shallow needling (0.30mm×25mm) at nonacupoints (located 1 inch beside acupoints).. Specifically, the depth of needle insertion into nonacupoints is 3-5mm and avoided manual stimulation and no "Deqi" without actual current output, and retained the needle for the same time as treatment group
  Arms: sham electroacupuncture treatment

SUMMARY:
1. Title: Effect of Electroacupuncture on Severe Acute Pancreatitis with Multiple Organ Disfunction Syndrome patients: A Randomized Clinical Trial
2. Research center: single center
3. Design of the research: A randomized, double-blind and parallel controlled study
4. Object of the research: The patients over 18 years that met the criteria of SAP and with more than 2 organs failure.
5. Sample size of the research: A total of 220patients,110 cases in each group
6. Interventions: The acupuncture points for electroacupuncture are Zusanli(ST36), Xiajuxu(ST39), Hegu(LI4), Neiguan(PC6) points . Participants in the treatment group underwent 30 minutes acupuncture (0.30mm×70mm) at above points once a day for seven days. After"Deqi",electroacupuncture stimulation apparatus (HANS G6805-2, Huayi Co, Shanghai, China) is connected and maintained the end of treatment. Participants in the control group received shallow needling (0.30mm×25mm) at nonacupoints (located 1 inch beside acupoints). Specifically, the depth of needle insertion into nonacupoints is 3-5mm and avoided manual stimulation and no "Deqi" without actual current output.
7. Aim of the research: To investigate the effect of electroacupuncture on Severe Acute Pancreatitis with Multiple Organ Disfunction Syndrome.
8. Outcome #Primary outcomes: All-cause 28-day mortality. Secondary outcomes: Duration of organ failure; The incidence of pancreatic necrotic tissue infection; Time for enteral nutrition to reach the standard (30kcal/kg); Mechanical ventilation time; Length of hospital stay
9. The estimated duration of the study#2 years.

DETAILED DESCRIPTION:
This study is a randomized, double-blinded, placebo controlled and long-term follow-up design. In this study, Zusanli(ST36), Xiajuxu(ST39), Hegu(LI4), Neiguan(PC6) were selected for electroacupuncture treatment, accompanied with evaluating the effects on 28-day mortality in SAP patients with MODS, as well as the duration of organ failure, the incidence of pancreatic necrotic tissue infection and length of hospital stay . To clarify the effect of electroacupuncture on SAP patients with MODS is of great significance to the clinical applications and popularization of traditional acupuncture treatment across the world.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnosis of severe acute pancreatitis (Atlanta diagnostic criteria), within 1 week of onset
2. Combine 2 or more organ failures at the same time, and the duration is greater than 48h
3. Age ≥18 years old;
4. Obtain informed consent.

Exclusion Criteria:

1. Pregnancy pancreatitis;
2. Patients who have undergone percutaneous puncture or surgical drainage before admission, and have undergone surgical decompression due to early abdominal hypertension;
3. Patients with a history of chronic organ dysfunction (such as uremia, COPD, liver cirrhosis, heart failure, etc.).
4. Those who have a medical history of acupuncture and moxibustion or are not sensitive to acupuncture and moxibustion.
5. Those who refuse to participate in the research

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-12-22 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
All-cause 28-day mortality | 1-2year
  All reasons (such as infection, hemorrhage) caused the mortality during the first 28 days after treatments

SECONDARY OUTCOMES:
Duration of organ failure | an average of 1-2 year
  The time of organ failure recovered
The incidence of pancreatic necrotic tissue infection | up to one year
  The incidence of pancreatic necrotic tissue infection
Duration of mechanical ventilation in patients with endotracheal intubation in ICU | an average of 1 year
  Duration of mechanical ventilation in patients with endotracheal intubation in ICU
Length of stay in hospital | 24 months
  ICU stay time and hospitalization time

REFERENCES:
- [Background] Bakker OJ, van Brunschot S, van Santvoort HC, Besselink MG, Bollen TL, Boermeester MA, Dejong CH, van Goor H, Bosscha K, Ahmed Ali U, Bouwense S, van Grevenstein WM, Heisterkamp J, Houdijk AP, Jansen JM, Karsten TM, Manusama ER, Nieuwenhuijs VB, Schaapherder AF, van der Schelling GP, Schwartz MP, Spanier BW, Tan A, Vecht J, Weusten BL, Witteman BJ, Akkermans LM, Bruno MJ, Dijkgraaf MG, van Ramshorst B, Gooszen HG; Dutch Pancreatitis Study Group. Early versus on-demand nasoenteric tube feeding in acute pancreatitis. N Engl J Med. 2014 Nov 20;371(21):1983-93. doi: 10.1056/NEJMoa1404393. PMID 25409371
- [Background] Kohli P, Gupta V, Kochhar R, Yadav TD, Sinha SK, Lal A. Lavage through percutaneous catheter drains in severe acute pancreatitis: Does it help?A randomized control trial. Pancreatology. 2019 Oct;19(7):929-934. doi: 10.1016/j.pan.2019.09.003. Epub 2019 Sep 9. PMID 31521496
- [Background] Karjula H, Nordblad Schmidt P, Makela J, Liisanantti JH, Ohtonen P, Saarela A. Prophylactic pancreatic duct stenting in severe acute necrotizing pancreatitis: a prospective randomized study. Endoscopy. 2019 Nov;51(11):1027-1034. doi: 10.1055/a-0865-1960. Epub 2019 Mar 20. PMID 30895583
- [Background] Liu Z, Yan S, Wu J, He L, Li N, Dong G, Fang J, Fu W, Fu L, Sun J, Wang L, Wang S, Yang J, Zhang H, Zhang J, Zhao J, Zhou W, Zhou Z, Ai Y, Zhou K, Liu J, Xu H, Cai Y, Liu B. Acupuncture for Chronic Severe Functional Constipation: A Randomized Trial. Ann Intern Med. 2016 Dec 6;165(11):761-769. doi: 10.7326/M15-3118. Epub 2016 Sep 13. PMID 27618593
- [Background] Liu Z, Liu Y, Xu H, He L, Chen Y, Fu L, Li N, Lu Y, Su T, Sun J, Wang J, Yue Z, Zhang W, Zhao J, Zhou Z, Wu J, Zhou K, Ai Y, Zhou J, Pang R, Wang Y, Qin Z, Yan S, Li H, Luo L, Liu B. Effect of Electroacupuncture on Urinary Leakage Among Women With Stress Urinary Incontinence: A Randomized Clinical Trial. JAMA. 2017 Jun 27;317(24):2493-2501. doi: 10.1001/jama.2017.7220. PMID 28655016